CLINICAL TRIAL: NCT05308264
Title: An Open-label, Phase 1b Study of R289, an IRAK1/4 Inhibitor, in Patients With Lower-risk Myelodysplastic Syndromes (LR MDS) Who Are Relapsed/Refractory/Resistant to Prior Therapies
Brief Title: Study of R289 in Patients With Lower-risk Myelodysplastic Syndromes (LR MDS)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C-906289-002
Record Dates: First submitted 2022-03-02; First posted 2022-04-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Low Risk Myelodysplastic Syndromes
Keywords: MDS; LR MDS; Myelodysplastic Syndromes; Hematology Oncology; Hem/ Onc
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): ESCALATION PHASE:
  Dose Level 1: 250mg PO qd Dose Level 2: 500mg PO qd Dose Level 3: 750 mg PO qd Dose Level 4: 250 mg PO bid Dose Level 5: 500 mg PO AM/250 mg PO PM Dose Level 6: 500 mg PO bid
  EXPANSION PHASE (randomized 1:1):
  Dose Level 1: 250 mg PO qd Dose Level 2: 250 mg PO bid
  Interventions: Drug: R906289 Monosodium (R289 Na)

INTERVENTIONS:
Drug: R906289 Monosodium (R289 Na) — Drug: R906289 Monosodium (R289 Na) R906289 Monosodium (250mg PO qd, 250mg PO bid, 500 mg PO qd, 500 mg PO bid, 750 mg PO qd, split dose - 500 mg PO AM/250 mg PO PM)
  Other Names: R906289 Monosodium

SUMMARY:
Phase 1b Study of R289 in Patients with Lower-risk Myelodysplastic Syndromes (LR MDS)

DETAILED DESCRIPTION:
An open-label, Phase 1b study of R289, an IRAK 1/4 Inhibitor, to determine tolerability and preliminary efficacy in patients with LR MDS who are relapsed/refractory/resistant, intolerant, or have inadequate response to prior therapies such as erythropoietin (EPO), luspatercept, or hypomethylating agents (HMAs) for MDS.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18 years of age at the time of signing the informed consent.
* Must have definitive diagnosis of MDS with very low, low, or intermediate-1 risk (International Prognostic Scoring System (IPSS)-R ≤ 3.5) and ≤5% bone marrow myeloblasts.
* Must be relapsed, refractory/resistant, intolerant, or have inadequate response to therapies with known clinical benefits for MDS, such as EPOs, luspatercept, and HMAs(i.e., azacytidine or decitabine). Patients with del (5q) must have failed prior lenalidomide therapy.
* DOSE ESCALATION PHASE:

  a. Must meet at least one of the following criteria prior to initial administration of study treatment: 1) Symptomatic anemia with hemoglobin < 9.0 g/dL and no RBC transfusion within 16 of registration or 2) RBC transfusion dependent defined as receiving ≥ 2 units of packed red blood cells (PRBCs) within 8 weeks in the preceding 16 weeks for a hemoglobin <9.0 g/dL.
* DOSE EXPANSION PHASE:

  1. Relapsed, refractory to or ineligible for ESAs and has previously received one or more approved therapies for LR-MDS
  2. Must be RBC transfusion dependent defined as receiving ≥ 2 units of packed red blood cells (PRBCs) within 8 weeks in the preceding 16 weeks for a hemoglobin <9.0 g/dL.
* EXPLORATORY PHASE 1b COHORT:

  1. Transfusion-dependent LR-MDS who are refractory or intolerant to, or are ineligible for ESAs.
  2. No prior therapy with any approved or investigational therapies for MDS
  3. No del 5q cytogenetic abnormality
  4. RBC transfusion dependent defined as receiving ≥ 2 units of PRBCs within 8 weeks in the preceding 16 weeks for a hemoglobin <9.0 g/dL
* All patients must have documented marrow iron stores. If marrow iron stain is not available, the transferrin saturation must be >20% or a serum ferritin > 100ng/100mL
* Must have Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2 at screening.
* Must have adequate organ function, defined as:

  1. Hepatic function:

     * aspartate amino transferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 × upper limit of normal (ULN)
     * total bilirubin ≤ 1.5 × ULN
  2. Renal function defined as creatinine clearance > 60 mL/min (using Cockcroft-Gault), or blood creatine < 1.5 mg/dL

Exclusion Criteria:

* Prior treatment for MDS (i.e., TPOs, EPOs, luspatercept, HMAs) concluded < 4 weeks prior to study treatment
* Clinically significant anemia resulting from iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis, or GI bleeding.
* MDS secondary to treatment with radiotherapy, chemotherapy, and/or immunotherapy for malignant or autoimmune diseases.
* Diagnosis of chronic myelomonocytic leukemia.
* History of uncontrolled seizures.
* Uncontrolled bacterial or viral infection (i.e., documented HIV, hepatitis B or hepatitis C).
* History of other malignancy that could affect compliance or interpretation of results. Patients with an malignancy other than leukemia appropriately treated with curative intent and the malignancy has been in remission without treatment for ≥ 2 years prior to study entry are eligible as are:

  1. Adequately treated in situ carcinoma of the cervix uteri
  2. Adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin, or
  3. Low grade, early-stage prostate cancer (Gleason score 6 or below, stage 1 or 2) with no requirement for therapy at any time prior to the study, or previously resected.
* History of or active, clinically significant, cardiovascular, respiratory, GI, renal, hepatic, neurological, psychiatric, musculoskeletal, genitourinary, dermatological, or other disorder that, in the Investigator's opinion (or following review by the Sponsor), could affect the conduct of the study or the absorption, metabolism or excretion of the study treatment.
* Prior history of autologous or allogeneic stem cell transplantation
* Marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval > 480 milliseconds [msec]) (Common Terminology Criteria for Adverse Events [CTCAE] Grade 1) using Fridericia's QT correction formula.
* History of additional risk factors for TdP (e.g., symptomatic heart failure with left ventricular ejection fraction [LVEF] <40%, hypokalemia, family history of Long QT Syndrome).
* Receiving any other concurrent chemotherapy, radiotherapy, or immunotherapy (within 2 weeks of initiating study treatment), or the toxicity of the relevant prior treatment has not been resolved yet. For any long-acting systemic agent such as a monoclonal antibody, study treatment should not begin within two half-lives of the agent.
* Use of concomitant medications that prolong the QT/QTc interval during study treatment
* Use of concomitant medications that are strong CYP3A or CYP2B6 inhibitors or inducers during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2 Year
  * Incidence of adverse events (AEs)
  * Incidence of discontinuation or interruptions of R289 due to AEs
  * Incidence of dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Outcome Measure: Preliminary Efficacy | 24 Weeks for Primary Efficacy; 8 Weeks for Characterized PK
  Measure Description Primary Efficacy:
  Proportion of patients achieving red blood cell transfusions independence by ≥ 8 weeks, ≥ 16 weeks, and ≥ 24 weeks Proportion of patients with overall response per IWG 2006 Proportion of patients with hematologic improvement per IWG 2018 Time Frame: 24 Weeks Measure Description Characterized PK Maximum plasma concentration (Cmax) Time Frame: 8 Weeks
Characterize pharmacokinetics (PK) | 8 Weeks
  Maximum plasma concentration (Cmax)

OTHER OUTCOMES:
Characterize pharmacodynamic (PD) | 1 year
  Change from baseline biomarker expression levels in plasma and bone marrow (including but not limited to, C-reactive protein [CRP] and tumor necrosis factor [TNF]-a)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - WashU Medicine, St Louis, Missouri
  - Oncology Clinical Research Referral Office, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Texas, Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Intermountain Healthcare, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No